CLINICAL TRIAL: NCT01400282
Title: Analgesic Efficacy of High Frequency Spinal Cord Stimulation: a Placebo-controlled Study
Brief Title: Analgesic Efficacy of High Frequency Spinal Cord Stimulation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ensemble Hospitalier de la Côte (Other)
Responsible Party: Perruchoud Christophe, MD, Ensemble Hospitalier de la Côte
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EHC-JCH
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-06

CONDITIONS: Lowback and Leg Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sequence 1 (Other): Conventional stimulation (2 weeks)- High frequeny stimulation (2 weeks)- Conventional stimulation (2 weeks)and sham stimulation (2 weeks)
  Interventions: Device: High frequency spinal cord stimulation
- Sequence 2 (Other): Conventional stimulation (2 weeks)- sham stimulation (2weeks) - Conventional stimulation (2 weeks) - high frequeny stimulation (2 weeks)
  Interventions: Device: High frequency spinal cord stimulation

INTERVENTIONS:
Device: High frequency spinal cord stimulation

SUMMARY:
The aim of the study is to compare the efficacy of high frequency (HF SCS) stimulation and sham stimulation (Sham SCS - i.e. no stimulation) and conventional spinal cord stimulation (Conv SCS) on the patient reported global impression of change, pain intensity and health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* treated with spinal cord stimulation
* stable pain relief achieved

Exclusion Criteria:

* failure to give informed consent
* unable to use or understand how to handle the equipment, PGIC,VAS score or EQ-5D questionnaires.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-06 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Patient's Global Impression of Change (PGIC)

SECONDARY OUTCOMES:
Intensity of Pain
Quality of Life (EQ-5D)

CONTACTS AND LOCATIONS:
Locations (2):
- Department of anesthesiology and Pain management, Ensemble Hospitalier de la Côte (EHC), Morges, Switzerland
- Department of Anaesthesia, The James Cook University Hospital, Middlesbrough, United Kingdom

REFERENCES:
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473